CLINICAL TRIAL: NCT01342874
Title: Improved Maternal and Fetal Outcomes Associated With Inositol Dietary Supplementation in Women With Early Gestational Diabetes Mellitus
Brief Title: Improved Outcomes Associated With Inositol Dietary Supplementation in Women With Gestational Diabetes Mellitus
Acronym: inositol
Status: Completed | Type: Observational
Sponsor: G. d'Annunzio University (Other)
Responsible Party: Principal Investigator, Claudio Celentano, MD, G. d'Annunzio University
Other Study IDs: INOS001
Record Dates: First submitted 2011-04-19; First posted 2011-04-27 (Estimated); Last update posted 2012-02-09 (Estimated); Status verified 2011-04

CONDITIONS: Gestational Diabetes Mellitus
Keywords: inositol; gestational diabetes mellitus; obstetric adverse outcomes
MeSH Terms: conditions — Diabetes, Gestational | interventions — Inositol

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Inositol group: Inositol dietary exposure 4000 mg/day
  Interventions: Dietary Supplement: Inositol
- Control group: folic acid 400 mcg/day

INTERVENTIONS:
Dietary Supplement: Inositol — inositol exposure in early GDM
  Groups: Inositol group

SUMMARY:
Objective: Insulin resistance during normal pregnancy and in gestational diabetes mellitus (GDM) are unknown. New criteria are based on fasting glucose levels since the beginning of pregnancy. Inositol, a putative second messenger of insulin, correlates with the degree of insulin resistance. Dietary supplementation of inositol improves insulin resistance in patients with GDM.

DETAILED DESCRIPTION:
Methods: A randomized double-blind study was carried out in women with GDM. Patients were randomly exposed to inositol and placebo. Increase of BMI, blood glucose at 75 grams oral glucose tolerance test (OGTT), fetal and neonatal adverse outcome, and insulin treatment were correlated to inositol exposure.

ELIGIBILITY:
Inclusion Criteria:

* singleton pregnant women
* random fasting glucose above 92 mg%

Exclusion Criteria:

* BMI >30
* random fasting glucose above 126 mg%

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: pregnant women presenting random fasting glucose during the first half of pregnancy above 92 mg%
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2010-08; Primary Completion 2011-04 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Insulin therapy in early diagnosis of GDM | 6 months
  Inositol supplementation and diet with/without insulin therapy in early GDM
altered OGTT | 6 months
  OGTT altered at 24-28 wks in inositol and control group

SECONDARY OUTCOMES:
delivery and neonatal outcomes | 6 months
  prevention of maternal and fetal adverse outcomes deriving from GDM (LGA fetuses, poly-hydramnios, C-section rate, gestational age at delivery, birthweight, birth injuries)

CONTACTS AND LOCATIONS:
Overall Officials: Claudio Celentano, MD, Principal Investigator — ObGyn Dept
Locations (1):
- University of Chieti, Chieti, CH, Italy

REFERENCES:
- [Background] Corrado F, D'Anna R, Di Vieste G, Giordano D, Pintaudi B, Santamaria A, Di Benedetto A. The effect of myoinositol supplementation on insulin resistance in patients with gestational diabetes. Diabet Med. 2011 Aug;28(8):972-5. doi: 10.1111/j.1464-5491.2011.03284.x. PMID 21414183